CLINICAL TRIAL: NCT05634356
Title: Social Influences on Sensorimotor Integration of Speech Production and Perception During Early Vocal Learning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Cornell University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Sarah Bottjer, Professor of Biology & Psychology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UP-18-00666; 1R21DC019773 (NIH)
Record Dates: First submitted 2022-11-04; First posted 2022-12-02 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Sensorineural Hearing Loss; Speech
MeSH Terms: conditions — Hearing Loss, Sensorineural; Speech

STUDY DESIGN:
Intervention Model Description: We have a parallel design in which parent-infant dyads are assigned to either the intervention or to a random control group.
Who Masked: Participant
Masking Description: Parents are not informed of their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Parents are instructed to say nonsense words in response to infant babbles with a conserved phonological form as infant plays.
  Interventions: Behavioral: vocal-social reinforcement
- Control (No Intervention): Parents are instructed to say nonsense words at random times with a conserved phonological form as infant plays.

INTERVENTIONS:
Behavioral: vocal-social reinforcement — experimental manipulation of social reinforcement in response to vocalizations
  Arms: Experimental

SUMMARY:
The goal of this study is to investigate the role of social factors on speech learning, including production and perception, in infants ranging in age from ~7-18 months. Infants have either typical hearing or sensorineural hearing loss. The main prediction of the study is that social reinforcement will engender improvements in vocal learning above and beyond gains in hearing in infants with hearing loss. As part of this study:

* The parent and infant engage in a free play session in the playroom while the investigator cues the parent to say simple nonsense words;
* Infants hear playback of the same words during a second phase.

DETAILED DESCRIPTION:
Infant vocal learning and development is embedded in a social feedback loop. Babbling vocalizations catalyze consistent responding by caregivers, and these predictable social reactions provide opportunities for infant learning. Naturalistic data and experimental manipulations have verified both the potency of babbling for eliciting social-vocal responses from caregivers, and the efficacy of social feedback for rapid advances in infant vocal learning. The impact of infant hearing loss, however, has never been studied with regard to the social feedback loop. Infants born with significant sensorineural hearing loss may be deprived not only of early auditory experience but of social experience as well. The reduction or elimination of social feedback to immature vocalizations, either by reduced or unpredictable parental responses or by infants' lessened ability to perceive those responses, is likely to have strong effects on learning and development of speech. Restoring hearing via cochlear implants improves auditory perception but does not remediate lost social learning opportunities or provide knowledge of how to learn from social partners. The goal of this project is to investigate how social interactions mediate the ability to incorporate phonological patterns of the language environment into vocal repertoires in infants with typical hearing versus infants with hearing loss (who either continue with hearing aids or experience gains in hearing via receipt of a cochlear implant). The investigators' method is to remotely observe naturally-occurring interactions between infants and a parent while recording their vocalizations; the investigators instruct the parent via headphones to provide vocal-social reinforcement to the infants when they produce a babbling utterance. Infant-parent dyads in a yoked control condition receive the same schedule of social reinforcement cues as a matched pair, which is random with respect to actual infant utterances in the control condition.

ELIGIBILITY:
Inclusion Criteria:

* infants ca. 7-16 months of age at study onset
* Infants less than 24 months of age (for follow-up visits only)
* At least one English-speaking or Spanish-speaking parent in the home who can participate in the study
* Subjects will include infants with typical hearing, hearing loss, or hearing loss remediated by a hearing aid or cochlear implant.

Exclusion Criteria:

* infants who are not exposed to English or Spanish in the home
* infants who do not have a parent who can participate in the study will be excluded (Caregivers who are not parents will not be eligible to participate in the study)

Ages: 7 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Vocal Codes During Study Visit | Measured over the course of 30 minutes
  Infant vocalizations are assigned to categories of speech maturity, and frequency of each category will be assessed before, during, and after the cued responses from parents.

SECONDARY OUTCOMES:
Change in Vocal Codes Between Visits | Measured at initial visit and up to three additional times between 30-180 days following the initial visit
  The same categories of speech maturity will be used at each study visit, allowing comparison of speech composition over time.
Perception | Measured at initial visit and up to three additional times between 30-180 days following the initial visit
  Infants will hear a recording of the same nonsense words spoken by their parent, and investigators will measure how long the infant looks in the direction of the word (how long the infant pays attention to each word).
MacArthur Communicative Development Inventory | assessed at 16 months and/or 6 months after initial visit
  This vocabulary inventory form will measure the breadth of the infant's known words and early sentence use.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah W Bottjer, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No